CLINICAL TRIAL: NCT01592149
Title: Survey of Prevalence of Loss of Appetite in Subject With Health Disorders.
Acronym: SPLASH
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16235
Record Dates: First submitted 2012-04-13; First posted 2012-05-07 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Appetite
Keywords: Appetite

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Other: No Drug

INTERVENTIONS:
Other: No Drug — No intervention will be given to subjects, survey of loss of appetite in patients suffering from various healthcare disorders.

SUMMARY:
The study is an epidemiological survey to find out the incidence of loss of appetite in Indian patients suffering from various health disorders. This survey will be conducted to obtain information on appetite from a total of 17500 subjects This study does not intend to study the effect of any drugs. The primary source of information will be the subjects themselves. The study will be conducted at 275 - 350 centres spread across India.This is a single visit study.The physician will conduct routine clinical, physical and general examination.

ELIGIBILITY:
Inclusion Criteria:

* Men and Non-pregnant women ≥ 18 years of age recuperating from healthcare disorders like:Malaria fever, Typhoid or enteric fever
* Hepatitis
* Acute infections including respiratory, urinary tract infections etc treated with antibiotic
* Tuberculosis
* Patient discharged from hospital after general surgical procedures like acute appendectomy, etc.
* Any other condition

Exclusion Criteria:

* Patients unwilling to provide informed consent & comply with the study procedure
* Patient using drugs which affect appetite like Cyproheptadine etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with various health related disoder
Sampling Method: Probability Sample
Enrollment: 16629 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with loss of appetite | 1 Day

SECONDARY OUTCOMES:
Percentage of patients with fatigue | 1 Day
Distribution of fatigue among the patients with respect to disease | 1 Day
Percentage of patients with moderate to very severe Fatigue. | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, India